CLINICAL TRIAL: NCT06036030
Title: Combination Momordica Charantia Extract and Primaquine Againts Plasmodium Falciparum Uncomplicated and Plasmodium Vivax Uncomplicated Treatment in Manokwari, West Papua
Acronym: MCMPFPB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syamsudin Abdillah,Ph.D, Pharm D (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other); PT Natura Nuswantara Nirmala (Unknown)
Responsible Party: Sponsor-Investigator, Syamsudin Abdillah,Ph.D, Pharm D, Profesor Dr Syamsudin Abdillah, M.Biomed, Pancasila University
Organization: Pancasila University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCMPFPB2019
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Malaria,Falciparum; Malaria, Vivax; Malaria; Infections; Uncomplicated Malaria; Uncomplicated Plasmodium Falciparum
Keywords: Momordica charantia; primaquine; combination therapy dihydroartemisinin; Plasmodium falciparum; Plasmodium vivax
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax; Malaria; Infections | interventions — artenimol; piperaquine; Primaquine; bitter melon extract

STUDY DESIGN:
Intervention Model Description: the patient comes to the primary health care facility, is examined by a doctor, if malaria is suspected, a parasite examination is carried out in the laboratory. If positive for falciparum malaria and based on the results of the doctor's examination meet the criteria as research subjects, then the drug is given based on the random table that has been provided.
Masking Description: The test drug and the control drug are put into the capsule with the same weight, type and smell so that the patient cannot distinguish between the test drug and the control drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bitter melon fruit extract (Momordica charantia) with primaquine (Experimental): For three days, a combination of 500 mg of bitter melon fruit extract (Momordica charantia) and 325 mg of bitter melon fruit content (13.50 mg/kg body weight) was administered. those with Plasmodium falciparum and Plasmodium vivax malaria received a single dosage of primaquine (0.25 mg/kg body weight) once daily, with those with Plasmodium falciparum malaria receiving it for 14 days.
  Interventions: Drug: Primaquine; Other: Momordica Charantia Extract
- dihydroartemisinin+piperaquine+ primaquine (Active Comparator): DHP (fixed dosage combination tablets containing 40 mg dihydroartemisinin and 320 mg piperaquine) was administered to the group for 3 days, with primaquine being administered for 14 days to patients with Plasmodium vivax and 1 day initially to those with Plasmodium falciparum without difficulties. Body weight is taken into consideration while setting therapy parameters (age 15 years, >40-60 kg: 3 tablets; >60-80 kg: 4 tablets; 80 kg: 5 tablets).
  Interventions: Drug: Dihydroartemisinin; Drug: Piperaquine; Drug: Primaquine

INTERVENTIONS:
Drug: Dihydroartemisinin — dihidroartemisinin dose of 2-4 mg/Kg Body weight taken for 3 days
  Arms: dihydroartemisinin+piperaquine+ primaquine
Drug: Piperaquine — piperaquine at a dose of 16-32 mg/Kg body weight taken for 3 days
  Arms: dihydroartemisinin+piperaquine+ primaquine
Drug: Primaquine — Primaquine dose 0.25 mg/kg body weight given to uncomplicated Plasmodium falciparum patients on the first day only
Other: Momordica Charantia Extract — Momordica charantia extract capsules at a dose of 325 mg were given to patients for 3 days
  Arms: bitter melon fruit extract (Momordica charantia) with primaquine

SUMMARY:
Comparing the efficacy of the combination treatment of bitter melon fruit extract (Momordica charantia) with primaquine (MC+PQ) against the combination of dihydroartemisinin + piperaquine + primaquine (DHP+PQ) on patients with Plasmodium falciparum and Plasmodium vivax without complications in Manokwari, West Papua, Indonesia. The research was conducted from January 2019 to April 2019 at Manokwari Regional General Hospital, West Papua. Open label, 2 parallel randomized clinical studies with Plasmodium falciparum malaria patients without complications (Study 1) and patients with Plasmodium vivax malaria without complications (Study 2). The randomized clinical trial divided in 2 treatment groups, namely the MC+PQ and DHP+PQ. The Success of the treatment was determined by the combination of blood schizontocidal therapy in radical cure. The overall final assessed results were the average value of parasitological failure, hematological measurements, liver function, kidney function, blood lipid levels, blood glucose levels and adverse events until day 42.

DETAILED DESCRIPTION:
Every group therapy session was under team member supervision, required to complete follow-up visits on days 1, 2, 3, 5, 7, 14, 21, 28, 35, and 42. All of the studies 1 and 2 was split into more than two treatment groups, MC+PQ and DHP+PQ. The study was broken up into several 2 studies. Plasmodium falciparum patients without complications (n = 50 in each study) were the subjects of study 1, and Plasmodium vivax patients without complications (n = 50) were the subjects of studies 2 and 3.

The combination of 500 mg of bitter melon fruit extract (Momordica charantia) and 325 mg of bitter melon fruit content (13.50 mg/kg body weight) was initially approved by the MC+PQ group and administered for 3 days. 15 mg Primaquine dose single (0.25 mg/kg body weight) was administered for patients with Plasmodium falciparum and Plasmodium vivax malaria. Patients with Plasmodium falciparum malaria was treated for the first 14 days, while those with Plasmodium vivax malaria were treated for 14 days.

The 2nd DHP+PQ group received three days of DHP (fixed dose combination tablets of 40 mg dihydroartemisinin and 320 mg piperaquine; DHP-FRIMAL, Mersi pharmaceutical, Tbk) in addition to 15 mg primaquine that had previously been given for one day to patients with Plasmodium falciparum who had no complications and for 14 days to those with Plasmodium vivax. DHP renewal is determined by body weight (age 15 years, >40-60 kg: 3 tablets; >60-80 kg: 4 tablets; 80 kg: 5 tablets)

ELIGIBILITY:
Inclusion Criteria:

* incomplete therapy patients
* Age ≥15 years old male or female up to 60 years old.
* diagnosis and an outcome inspection microscopically suffering from Plasmodium falciparum malaria or Plasmodium vivax with density parasites 1000-100,000/µL
* History of fever within the past 24-48 hours with axillary temperature ≥ 37.5°C
* There were no signs of severe malaria
* had no chronic disease
* willing to follow up for 42 days; No consuming other antimalarial drugs within 2 weeks; willingly to participate in investigations and follow established procedures (informed consent)

Exclusion Criteria:

* pregnant female, breastfeeding female, children and infants
* suffering a mental disturbance, heavy illness like kidney, liver, tuberculosis, cancer, AIDS and other heavy diseases
* one set of symptom or signs of severe malaria
* had a history of hypersensitivity, allergies, and antimalarial contraindications
* not willingly to follow the inquiry

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
development of sexual and asexual stages of Plasmodium falciparum | 0, 14, 28, and 42 days post-treatment
  Finger prick blood samples are collected for malaria blood smear. Thick and thin blood smear were stained with 3% giemsa solution for 45 minutes and were read under binocular microscope with 1,000x magnification

SECONDARY OUTCOMES:
Parasite clearence times | 0, 14, 28, and 42 days post-treatment
  parasite reduction ratio
Fever clearance time | 0, 14, 28, and 42 days post-treatment
  time taken for the axilla temperature to fall below 37.5°C in patients who were febrile at inclusion

OTHER OUTCOMES:
Hemoglobin measurement | 0, 14, 28, and 42 days post-treatment
  Hematological study, measure in g/dl
Erytrocytes measurement | 0, 14, 28, and 42 days post-treatment
  Hematological study, measure in 10^6/mm³
Hematocrits measurement | 0, 14, 28, and 42 days post-treatment
  Hematological study, measure in %
Thrombocytes measurement | 0, 14, 28, and 42 days post-treatment
  Hematological study, measure in 10^3/mm³
Leucocytes measurement | 0, 14, 28, and 42 days post-treatment
  Hematological study, measure count in 1 µL
Albumin measurement | 0, 14, 28, and 42 days post-treatment
  Hematological study, measure in mg%
AST/SGOT measurement | 0, 14, 28, and 42 days post-treatment
  Blood chemistry, measure in µ/mL
total bilirubin measurement | 0, 14, 28, and 42 days post-treatment
  Blood chemistry, measure in mg %
Direct bilirubin measurement | 0, 14, 28, and 42 days post-treatment
  Blood chemistry, measure in mg %
Total protein measurement | 0, 14, 28, and 42 days post-treatment
  Blood chemistry, measure in mg %
Creatinine measurement | 0, 14, 28, and 42 days post-treatment
  Blood chemistry, measure in mg %
Ureum measurement | 0, 14, 28, and 42 days post-treatment
  Blood chemistry, measure in mg %
Gout measurement | 0, 14, 28, and 42 days post-treatment
  Blood chemistry, measure in mg %
Total Cholesterol measurement | 0, 14, 28, and 42 days post-treatment
  Lipid parameter, measure in mg/dL
Triglycerides measurement | 0, 14, 28, and 42 days post-treatment
  Lipid parameter, measure in mg/dL
Glucose measurement | 0, 14, 28, and 42 days post-treatment
  Glucose parameter, measure in mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Manokwari Regional General Hospital, Manokwari, West Papua, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year
Access Criteria: Sharing Access are only for research purposes.

REFERENCES:
- [Background] Abdillah S, Tambunan RM, Sinaga YM, Farida Y. Ethno-botanical survey of plants used in the traditional treatment of malaria in Sei Kepayang, Asahan of North Sumatera. Asian Pac J Trop Med. 2014 Sep;7S1:S104-7. doi: 10.1016/S1995-7645(14)60213-3. PMID 25312101
- [Background] Jia S, Shen M, Zhang F, Xie J. Recent Advances in Momordica charantia: Functional Components and Biological Activities. Int J Mol Sci. 2017 Nov 28;18(12):2555. doi: 10.3390/ijms18122555. PMID 29182587
- [Background] Chen F, Huang G, Yang Z, Hou Y. Antioxidant activity of Momordica charantia polysaccharide and its derivatives. Int J Biol Macromol. 2019 Oct 1;138:673-680. doi: 10.1016/j.ijbiomac.2019.07.129. Epub 2019 Jul 22. PMID 31344411
- [Background] Wang S, Liu Q, Zeng T, Zhan J, Zhao H, Ho CT, Xiao Y, Li S. Immunomodulatory effects and associated mechanisms of Momordica charantia and its phytochemicals. Food Funct. 2022 Nov 28;13(23):11986-11998. doi: 10.1039/d2fo02096c. PMID 36350105
- [Result] Nelwan EJ, Ekawati LL, Tjahjono B, Setiabudy R, Sutanto I, Chand K, Ekasari T, Djoko D, Basri H, Taylor WR, Duparc S, Subekti D, Elyazar I, Noviyanti R, Sudoyo H, Baird JK. Randomized trial of primaquine hypnozoitocidal efficacy when administered with artemisinin-combined blood schizontocides for radical cure of Plasmodium vivax in Indonesia. BMC Med. 2015 Dec 11;13:294. doi: 10.1186/s12916-015-0535-9. PMID 26654101